

# **Title Page**

Protocol Title: A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of AGN-190584 in Participants

with Presbyopia

**Protocol Number: 1883-301-013** 

**Amendment Number: 1** 

Product: AGN-190584

**Brief Protocol Title:** Phase 3 efficacy study of AGN-190584 in participants with presbyopia

**Development Phase: 3** 

Sponsor Name: Allergan, Inc.

**Legal Registered Address:** 

2525 Dupont Drive, Irvine, CA 92612, USA

**Serious Adverse Event Reporting:** 

**Allergan Medical Safety Physician Contact Information:** 

#### **Allergan Signatory:**

Vice President, Therapeutic Area Head Anterior Segment and Consumer Eye Care Allergan, Inc.

Refer to the final page of this protocol for electronic signature and date of approval.



# **Protocol Amendment Summary of Changes**

| DOCUMENT HISTORY | |
|-------------------|------------------|
| Document | Date |
| Amendment 1 | 05 December 2018 |
| Original Protocol | 13 October 2018 |

# Amendment 1 (05 December 2018)

#### **Overall Rationale for the Amendment:**

The following is a summary of changes made to the original protocol, some of which are based on communication with the FDA.

| Section No. and<br>Name | Description of Change | Brief Rationale |
|---|---|---|
| Throughout | Update figures, tables, appendices, and text to a 30-day study intervention timeline | A 30-day study intervention period is an adequate duration to demonstrate safety and efficacy of AGN-190584 |
| 1.1. Synopsis; 1.3. Schedule of Activities; 3. Objectives and Endpoints; 8. Study Assessments and Procedures; 10.7. Appendix 7 | Add OD and OS measurements for mesopic and photopic CDVA, DCIVA, and DCNVA | In addition to binocular measurements, individual eye measurements were added to mesopic and photopic CDVA, DCIVA, and DCNVA to provide a more complete assessment of these endpoints |
| 1.1. Synopsis; 4.1. Overall Design; 9.2. Sample Size Determination | Modify participant dropout rate to 10% and participants completing the study per study intervention group to approximately 135 | The participant dropout rate assumption was modified to 10% (versus 20%) as this is a sufficiently conservative estimate of participants who may not complete the 30-day study. Assumptions for the sample size calculation and their basis were clarified. |
| 1.1. Synopsis; 6.3. Measures to Minimize Bias: Randomization and Blinding; 9.4.1.3. Secondary Analyses; 9.4.4.1. Subgroup Analyses | Modify "baseline DCNVA" to "baseline binocular DCNVA" for randomization and analysis | "Baseline DCNVA" was modified to "baseline<br>binocular DCNVA" to clarify this stratification<br>parameter during randomization and statistical<br>analysis |
| 1.3. Schedule of<br>Activities; 8.8.<br>Biomarkers and<br>Other | Add determination of dominant eye | Collection of participant dominant/nondominant eye data was clarified |



| Section No. and<br>Name | Description of Change | Brief Rationale |
|---|---|---|
| Assessments; 10.7. Appendix 7 | | |
| 1.3. Schedule of<br>Activities; 10.7.1.<br>Screening Visit<br>(Days -30 to -1) | Modify screening DCNVA assessment that will be repeated 3 times with different charts to OD only | OD was added to clarify that the screening visit DCNVA (to be repeated 3 times with different charts) is for OD only |
| 7.1. Discontinuation of Study Intervention | Added a guideline to encourage participants who discontinue the study intervention early to stay in the study for the safety assessments at Day 30 | This was added to promote a continuation of safety assessments if a participant discontinues study intervention before the end of the study |
| 9.1. Statistical<br>Hypotheses | Update of statistical hypotheses | The statistical hypotheses for the primary and key secondary efficacy endpoints were clarified |
| 9.2. Sample Size<br>Determination | Update of sample size justification | The vehicle group intervention effect was updated based on previous phase 2 study results; the intervention effect for the non-emmetropes group was added. The total number of participants to complete the study was changed to 135 for each treatment group |
| 9.4.1. Efficacy<br>Analyses | Remove key secondary efficacy endpoint (change from baseline letters AUC <sub>0-10</sub> in mesopic, high contrast, binocular DCNVA at Day 30) and its analysis method | This key secondary efficacy endpoint is not required to demonstrate the efficacy of AGN-190584 |
| 9.4.1.1. Analysis<br>Endpoints | Remove secondary efficacy endpoint (photopic, high contrast, binocular DCIVA mean change from baseline letters AUC <sub>0-10</sub> at Day 30) and its analysis method | This secondary efficacy endpoint is not required to demonstrate the efficacy of AGN-190584 |
| 9.4.1.1. Analysis<br>Endpoints | Add secondary efficacy endpoint<br>(Change from baseline photopic, high<br>contrast, binocular DCIVA letters at<br>Day 30, Hour 3) | This secondary efficacy endpoint was added to evaluate the efficacy of AGN-190584 for DCIVA |
| 9.4.1.3.<br>Secondary<br>Analyses | Update change from baseline analysis (MMRM) | The change from baseline analysis model (MMRM) was updated to include the following additional fixed effects: visit, visit by study intervention group interaction, and baseline value by visit interaction |
| 9.4.4.1 Subgroup<br>Analyses | Update subgroup analyses | Subgroup analyses by gender and race was added |
| Throughout | Minor editorial and document formatting revisions | Minor, therefore have not been summarized |



# **Table of Contents**

| | ol Amendment Summary of Changes | |
|---------|-------------------------------------------------------|----|
| | of Contents | |
| List of | Tables | 7 |
| List of | Figures | 7 |
| 1. | Protocol Summary | 8 |
| 1.1. | Synopsis | |
| 1.2. | Schema | 10 |
| 1.3. | Schedule of Activities | 11 |
| 2. | Introduction | 18 |
| 2.1. | Study Rationale | |
| 2.2. | Background | 18 |
| 2.3. | Benefit/Risk Assessment | 19 |
| 3. | Objectives and Endpoints | 20 |
| 4. | Study Design | |
| 4.1. | Overall Design | |
| 4.1.1. | Clinical Hypotheses | |
| 4.2. | Scientific Rationale for Study Design | |
| 4.3. | Justification for Dose | |
| 4.4. | End of Study Definition | |
| 5. | Study Population | 23 |
| 5.1. | Inclusion Criteria | |
| 5.2. | Exclusion Criteria | |
| 5.3. | Lifestyle Considerations | 26 |
| 5.4. | Screen Failures | |
| 6. | Study Intervention | 27 |
| 6.1. | Study Intervention(s) Administered | 27 |
| 6.1.1. | Study Supplies | |
| 6.1.2. | Instructions for Use and Administration | 28 |
| 6.2. | Preparation/Handling/Storage/Accountability | 28 |
| 6.3. | Measures to Minimize Bias: Randomization and Blinding | 29 |
| 6.4. | Study Intervention Compliance | |
| 6.5. | Concomitant Therapy | |
| 6.5.1. | Prohibited Interventions and Washout Before the Study | 30 |
| 6.5.2. | Permitted Interventions | |
| 6.5.3. | Rescue Medicine | |
| 6.5.4. | Prohibited Interventions During the Study | 31 |



| AGN-1 | 90584 | |
|---|---|---|
| 6.6. | Dose Modification | 31 |
| 6.7. | Intervention after the End of the Study | 31 |
| 7. | Discontinuation of Study Intervention and Participant | |
| <b>/•</b> | Discontinuation/Withdrawal | 32 |
| 7.1. | Discontinuation of Study Intervention | |
| 7.2. | Participant Discontinuation/Withdrawal from the Study | |
| 7.3. | Lost to Follow Up | |
| 8. | Study Assessments and Procedures | 34 |
| 8.1. | Efficacy Assessments | |
| 8.2. | Safety Assessments | |
| 8.2.1. | Vital Signs | |
| 8.2.2. | Pregnancy Testing. | |
| 8.2.3. | Photopic and Mesopic, High Contrast Corrected Distance Visual | |
| | Acuity for Each Eye and Binocularly | 38 |
| 8.2.4. | Near Contrast Sensitivity | |
| 8.2.5. | Study Intervention Tolerability and Drop Comfort Assessments | 38 |
| 8.2.6. | Temporal/Supraorbital Headache Visual Analog Scale | 38 |
| 8.2.7. | Intraocular Pressure | |
| 8.2.8. | Slit-lamp Biomicroscopy | 39 |
| 8.2.9. | Manifest Refraction | 42 |
| 8.2.10. | Dilated Funduscopic Examination | 42 |
| 8.2.11. | Suicidal Risk Monitoring | 43 |
| 8.3. | Adverse Events and Serious Adverse Events | 43 |
| 8.3.1. | Time Period and Frequency for Collecting Adverse Event and | |
| | Serious Adverse Event Information | 43 |
| 8.3.2. | Method of Detecting Adverse Events and Serious Adverse | |
| | Events | |
| 8.3.3. | Follow-up of Adverse Events and Serious Adverse Events | |
| 8.3.4. | Regulatory Reporting Requirements for Serious Adverse Events | |
| 8.3.5. | Pregnancy | |
| 8.3.6. | Medication Errors | |
| 8.4. | Treatment of Overdose | |
| 8.5. | Pharmacokinetics | |
| 8.5.1. | Blood Pharmacokinetic Sampling Procedure | |
| 8.5.2. | Pharmacokinetic Sample Bioanalysis | |
| 8.6. | Pharmacodynamics | |
| 8.7. | Genetics | |
| 8.8. | Biomarkers and Other Assessments | |
| 8.8.1. | Biomarkers | |
| 8.8.2. | Determination of Dominant Eye | |
| 8.9. | Health Economics | 48 |
| 9. | Statistical Considerations | 48 |



| ٨ | GN | $J_{\perp}^{1}$ | l Qí | 158 | 1 |
|---|----|-----------------|------|-----|---|

| 9.1. | Statistical Hypotheses | 48 |
|---|---|---|
| 9.2. | Sample Size Determination | |
| 9.3. | Populations for Analyses | |
| 9.4. | Statistical Analyses | |
| 9.4.1. | Efficacy Analyses | |
| 9.4.2. | Safety Analyses | |
| 9.4.3. | Pharmacokinetic Analyses | |
| 9.4.4. | Other Analyses | |
| 9.5. | Interim Analyses | 53 |
| 9.5.1. | Data Monitoring Committee | |
| 10. | Supporting Documentation and Operational Considerations | <b>5</b> 4 |
| 10.1. | Appendix 1: Regulatory, Ethical, and Study Oversight | |
| | Considerations | |
| 10.1.1. | Regulatory and Ethical Considerations. | |
| 10.1.2. | Financial Disclosure | |
| 10.1.3. | Informed Consent Process | |
| 10.1.4. | Data Protection. | 56 |
| 10.1.5. | Posting Clinical Study Data | |
| 10.1.6. | Data Quality Assurance | |
| 10.1.7. | Source Documents | |
| 10.1.8. | Study and Site Closure | |
| 10.1.9. | Publication Policy | |
| 10.1.10. | Compliance with Protocol. | 58 |
| 10.2. | Appendix 2: Adverse Events: Definitions and Procedures for | |
| | Recording, Evaluating, Follow-up, and Reporting | |
| | on of AE | |
| Definition | on of SAE | 60 |
| | ng and Follow-Up of AEs and/or SAEs | |
| - | ng of SAEs | |
| 10.3. | Appendix 3: Abbreviations | |
| 10.4. | Appendix 4: Standard Discontinuation Criteria | 66 |
| 10.5. | Appendix 5: Study Tabular Summary | 68 |
| 10.6. | Appendix 6: Contraceptive Guidance and Collection of | |
| | Pregnancy Information | 70 |
| | ons: | |
| | eption Guidance: | |
| | cy Testing: | |
| Collection | on of Pregnancy Information: | 72 |



| 10.8. | Appendix 8: Patient Reported Outcomes Questionnaires, |
|----------|---------------------------------------------------------|
| 10.0. | Descriptions, and Instructions |
| 10.8.1. | National Eye Institute Visual Function Questionnaire 25 |
| 10.8.2. | Near Vision Presbyopia Task-based Questionnaire |
| 10.8.3. | Presbyopia Impact and Coping Questionnaire |
| 10.8.4. | Presbyopia Patient Satisfaction Questionnaire |
| 10.8.5. | Patient Global Impression of Status |
| 10.8.6. | Patient Global Impression of Change |
| 10.8.7. | Patient Expectations for Treatment Efficacy |
| 11. | References 125 |
| | List of Tables |
| Table 1- | |
| Table 1- | Schedule of Visits and Procedures: Screening to Visit 3 |
| | Schedule of Visits and Procedures: Screening to Visit 3 |
| Table 1- | Schedule of Visits and Procedures: Screening to Visit 3 |
| Table 1- | Schedule of Visits and Procedures: Screening to Visit 3 |



# 1. Protocol Summary

## 1.1. Synopsis

**Protocol Title:** A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of AGN-190584 in Participants with Presbyopia

**Protocol Number:** 1883-301-013

**Brief Title:** Phase 3 efficacy study of AGN-190584 in participants with presbyopia

#### **Study Rationale:**

In previous studies, Allergan established the safety and efficacy of several (0.5% to 1.5%) concentrations of AGN-190584 dosed once daily, bilaterally or in the nondominant eye, over a period of up to 28 days in participants with presbyopia. Study 1883-301-013 is a multicenter, double-masked, randomized, vehicle-controlled, parallel group, Phase 3 study evaluating the efficacy, safety, and pharmacokinetics of AGN-190584 (1.25% pilocarpine) dosed once daily, bilaterally, over a period of 30 days in participants with presbyopia.

#### **Objectives and Measures:**

The objectives of this study are to evaluate the efficacy, safety, and pharmacokinetics of AGN-190584 when administered bilaterally, once daily for 30 days in participants with presbyopia.



| Objectives | Measures |
|---|---|
| To evaluate the efficacy of AGN-190584 when administered bilaterally, once daily for 30 days in participants with presbyopia. | <ul> <li>Mesopic and photopic, high contrast distance-corrected near visual acuity (DCNVA) for each eye and binocularly</li> <li>Mesopic and photopic, high contrast distance-corrected intermediate visual acuity for each eye and binocularly</li> <li>Patient reported outcomes questionnaires: <ul> <li>Mesopic and Photopic Near Vision Presbyopia Taskbased Questionnaire</li> <li>Presbyopia Impact and Coping Questionnaire</li> </ul> </li> </ul> |
| To evaluate the safety and tolerability of AGN-190584 when administered bilaterally, once daily for 30 days in participants with presbyopia | <ul> <li>Adverse events</li> <li>Photopic and mesopic high contrast corrected distance visual acuity for each eye and binocularly</li> <li>Near Contrast sensitivity</li> <li>Vital signs (blood pressure and heart rate)</li> <li>Study drug tolerability and drop comfort assessments</li> <li>Temporal/supraorbital headache visual analog scale</li> <li>Intraocular pressure</li> <li>Slit-lamp biomicroscopy</li> <li>Manifest refraction</li> <li>Dilated funduscopic examination</li> <li>Pregnancy test for women of childbearing potential</li> </ul> |
| To evaluate the pharmacokinetics of AGN-190584 when administered bilaterally, once daily for 30 days in participants with presbyopia | Plasma concentrations of AGN-190584 (sampled at selected sites; approximately 10% of all enrolled participants) |

#### **Overall Study Design:**

This is a multicenter, double-masked, randomized, parallel-group, vehicle-controlled, Phase 3 study in participants with presbyopia. The study population will consist of adult male and female participants with objective and subjective evidence of presbyopia.

#### **Number of Participants:**

Approximately 150 participants per group will be enrolled to achieve at least 135 participants per group completing the study based on an assumed dropout rate of 10%. Participants who prematurely discontinue from the study will not be replaced.



#### **Number of Sites:**

There will be approximately 50 sites in the United States.

#### **Intervention Groups and Study Duration:**

Participants will be randomized in a 1:1 ratio to receive either AGN-190584 or vehicle dosed once daily, in each eye, for 30 days. This randomization will be stratified by age (2 groups:  $\leq$  50 years and  $\geq$  50 years), baseline binocular DCNVA (2 groups: 20/40 to 20/60 inclusively, and worse than 20/60), iris color (brown and non-brown), and emmetropes/non-emmetropes. This study consists of the following visits: screening (Days -30 to -1), Day 1 (baseline), and Days 3, 7, 14, and 30.

#### **Data Monitoring Committee:** No

#### 1.2. Schema

The study schema is provided in Figure 1-1.

Figure 1-1 Study Schema



# 1.3. Schedule of Activities















Table 1–2 Schedule of Visits and Procedures: Visit 4 to Visit 5/Early Exit









#### 2. Introduction

Allergan is investigating pilocarpine HCl ophthalmic solution 1.25% (AGN-190584) as a noninvasive, reversible, pharmacological treatment for presbyopia, a condition in which the eye exhibits a diminished ability to focus on near objects with increasing age.

## 2.1. Study Rationale

In previous studies, Allergan established the safety and efficacy of various concentrations of AGN-190584 dosed once daily, bilaterally or in the nondominant eye, over a period of up to 28 days in participants with presbyopia. Study 1883-301-013 is a multicenter, double-masked, randomized, vehicle-controlled, parallel group, Phase 3 study evaluating the safety, efficacy, and tolerability of AGN-190584 dosed once daily, bilaterally, over a period of 30 days in participants with presbyopia.

# 2.2. Background

The impairment of near vision is common among older adults. In 2005, 1.044 billion people globally were estimated to have presbyopia, and prevalence is expected to increase to 1.782 billion by 2050 (Holden 2008). Both nonsurgical and surgical methods for the correction of presbyopia are available. Traditional nonsurgical methods of refractive correction for presbyopia include the use of dedicated reading spectacles, bifocal or varifocal spectacles, and monovision or multifocal contact lenses. A number of surgical techniques are also used for the treatment of presbyopia, which include monovision PRK or LASIK, conductive keratoplasty, intraocular lenses, and corneal inlays. However, for each of the existing technologies mentioned above, visual quality is reduced at 1 or more viewing distances, and each comes with its own unique safety risks and associated complications. For example, bifocals and progressive lenses (eg. reading glasses, contacts) produce optical aberrations and can increase the risk of falls (Johnson 2007, Lord 2002). Multifocal optics reduce image quality uniformly at all viewing distances. For surgical technologies, surgical risks, and the need for repositioning and explantation, or regression of effect have limited their widespread adoption (Moshirfar 2017, Ruiz 2009, Tomita 2015). Thus, there remains a need for a noninvasive, reversible, pharmacological treatment for presbyopia.

Pilocarpine is a muscarinic receptor agonist that mimics the actions of the parasympathetic neurotransmitter, acetylcholine, on smooth muscle. This causes 2 effects that enhance near vision: 1) constriction of the iris sphincter muscle, resulting in pupil constriction (miosis), and 2) contraction of the ciliary muscle, resulting in central lens steepening and lens accommodation (focusing from distance to near) (García-Lázaro 2012). Reducing the pupil size has long been recognized as an effective way to increase the useful depth of focus, in part by reducing peripheral aberrations (Tucker 1975).

Pilocarpine ophthalmic solutions are currently used for the reduction of elevated IOP in patients with open-angle glaucoma or ocular hypertension, management of acute-angle closure glaucoma,



prevention of postoperative elevated IOP associated with laser surgery, and induction of miosis (Pilocarpine HCl ophthalmic solution package insert 2011). Currently, the use of pilocarpine ophthalmic solution is limited by the commonly experienced AE of temporal and periorbital headache (ie, brow ache), which is believed to be due to the rapidity of the ciliary muscle contraction (Tsai 2009). However, Allergan has established an acceptable safety profile of AGN-190584 in 3 Phase 2 clinical studies (Studies 199201-007, 199201-009, and 199201-010). This is likely because the posology of pilocarpine evaluated for the treatment of presbyopia to date is of lower concentration (0.5% to 1.5%) and less frequently administered (once to twice daily) than for the treatment of glaucoma (1.0% to 4.0% administered up to 4 times daily). As a result, discontinuation rates for all Phase 2 clinical studies were generally low and safety parameters were not clinically significant between participants that received AGN-190584 compared to participants that received vehicle or a combination therapy. The majority of AEs reported in any treatment group were mild to moderate in intensity.

Efficacy measures for Phase 2 clinical studies included mesopic uncorrected near visual acuity line and letter improvement. Of the various concentrations of AGN-190584 evaluated, near vision was most improved compared with vehicle under mesopic and photopic conditions at the 1.0% and 1.5% pilocarpine concentrations, respectively.

More detailed information regarding clinical safety findings, clinical efficacy findings, chemistry, and pharmacology is provided in the IB.

#### 2.3. Benefit/Risk Assessment

Currently available approaches to presbyopia correction include nonsurgical options (spectacles or contact lenses) and surgical options (PRK or LASIK, conductive keratoplasty, intraocular lenses, or corneal inlays). Each approach has its own risk-benefit ratio. Because the risk-benefit ratio with nonsurgical options is generally lower than that of surgical procedures, both historical and contemporary practice has been to attempt nonsurgical or pharmacological treatment before resorting to more invasive alternatives.

Although the use of spectacles and contact lenses to correct presbyopia is widespread, this approach has limitations. Multifocal spectacles impair depth perception and edge-contrast sensitivity at critical distances for detecting obstacles in the environment (Lord 2002), and varifocal lenses have a corridor of nondistorted vision. For these reasons, older people are more than twice as likely to fall when wearing multifocal spectacles, and many participants have difficulty adjusting to using them (Johnson 2007, Lord 2002). As a result, Allergan is developing a noninvasive, reversible, pharmacological treatment for presbyopia.

More detailed information about the known and expected benefits and risks and reasonably expected AEs of AGN-190584 may be found in the IB.



# 3. Objectives and Endpoints

| Objectives | Measures |
|---|---|
| To evaluate the efficacy of AGN-190584 when administered bilaterally, once daily for | Mesopic and photopic, high contrast DCNVA for each eye and binocularly |
| 30 days in participants with presbyopia. | • Mesopic and photopic, high contrast DCIVA for each eye and binocularly |
| | PRO questionnaires: |
| | <ul> <li>Mesopic and Photopic NVPTQ</li> </ul> |
| | o PICQ |
| To evaluate the safety and tolerability of | • AEs |
| AGN-190584 when administered bilaterally, | <ul> <li>Photopic and mesopic high contrast CDVA for each eye</li> </ul> |
| once daily for 30 days in participants with presbyopia | and binocularly |
| | Near Contrast sensitivity |
| | • Vital signs (blood pressure and heart rate) |
| | Study drug tolerability and drop comfort assessments |
| | Temporal/supraorbital headache VAS |
| | • IOP |
| | Slit-lamp biomicroscopy |
| | Manifest refraction |
| | Dilated funduscopic examination |
| | <ul> <li>Pregnancy test for WOCBP</li> </ul> |
| To evaluate the pharmacokinetics of AGN-190584 when administered bilaterally, once daily for 30 days in participants with presbyopia | Plasma concentrations of AGN-190584 (sampled at selected sites; approximately 10% of all enrolled participants) |



## 4. Study Design

# 4.1. Overall Design

This is a multicenter, double-masked, randomized, parallel-group, vehicle-controlled, Phase 3 study in participants with presbyopia. Participants will receive AGN-190584 or vehicle dosed once daily, bilaterally, for 30 days. Approximately 300 participants with presbyopia will be enrolled at approximately 50 sites in the United States.

This study consists of the following visits: screening, Day 1 (baseline), and Days 3, 7, 14, and 30. A study schema is located in Section 1.2 and the SoA is located in Section 1.3.

Approximately 150 participants per group will be enrolled to achieve at least 135 participants per group completing the study. Participants who prematurely discontinue from the study will not be replaced.

#### 4.1.1. Clinical Hypotheses

- AGN-190584 ophthalmic solution dosed bilaterally, once daily for 30 days will demonstrate a significant improvement in DCNVA over vehicle.
- AGN-190584 ophthalmic solution dosed bilaterally, once daily for 30 days will demonstrate an acceptable safety and tolerability profile.

# 4.2. Scientific Rationale for Study Design

The current Phase 3 clinical study is designed to evaluate the efficacy, safety, and tolerability of AGN-190584 versus vehicle over a 30-day study intervention period when administered once daily bilaterally in participants with presbyopia.

Allergan Phase 2 Studies 199201-007 and 199201-009 support the administration of AGN-190584 monotherapy as an effective and safe treatment for presbyopia in doses up to 1.5%. The current Phase 3 study will evaluate AGN-190584 in an expanded participant population to establish efficacy and safety.

#### 4.3. Justification for Dose

Through modeling and evaluation of the Phase 2 results (Studies 199201-007, 199201-009, and 199201-010), Allergan has determined the optimal dose of AGN-190584 to be 1.25% for the treatment of presbyopia.

# 4.4. End of Study Definition

The EOS is defined as the date of the last visit of the last participant in the study.



A participant is considered to have completed the study if he/she has completed all phases of the study including the last visit.



# 5. Study Population

The study population will consist of adult male and female participants with objective and subjective evidence of presbyopia.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

## 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

| 1. | Age |
|---|---|
| 1.01 | Participant must be 40 to 55 years of age inclusive, at the time of the screening visit |
| 2. | Type of Participant and Presbyopia Characteristics |
| 2.01 | In good general health at the screening visit, as determined by the investigator |
| 2.02 | Subjective complaints of poor near vision that impact activities of daily living, |
| 3. | Sex |



| 3.01 | Male and female |
|---|---|
| 4. | Informed Consent |
| 4.01 | Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol |
| 4.02 | Written informed consent from the participant or a legally authorized representative has been obtained prior to any study-related procedures |
| 4.03 | Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information for the United States) |
| 5. | Other |
| 5.01 | Able, as assessed by the investigator, and willing to follow study instructions and likely to complete all required study visits |

# 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

| 1. | Medical Conditions |
|---|---|
| 1.01 | Uncontrolled systemic disease |
| 1.03 | Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of AGN-190584. History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery, radial keratotomy, or any intraocular surgery. However, participants with history of PRK or LASIK with CDVA meeting inclusion criteria will be allowed to enroll. |
| 1.04 | Known allergy or sensitivity to the study intervention or its components or other cholinergic agonist medications |
| 2. | Prior/Concomitant Therapy |



| 2.01 | Concurrent use of any topical ophthalmic medications, including artificial tears, other than the study intervention during the course of the study |
|---|---|
| 2.02 | Concurrent use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes |
| 3. | Prior/Concurrent Clinical Study Experience |
| 3.01 | Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study |
| 3.02 | Participation in a blood or plasma donation program within 30 days prior to study intervention administration |
| 4. | Diagnostic Assessments |
| 4.02 | Severe dry eye disease (defined as total corneal staining $\geq$ grade 3 on the 5-point Oxford scale and an OSDI score of $>$ 33) at the screening visit |
| 4.03 | Corneal abnormalities (including keratoconus, corneal scar, Fuchs' endothelial dystrophy, guttata, or edema) in either eye that are likely to interfere with visual acuity |
| 4.04 | Narrow iridocorneal angles (Shaffer grade ≤ 2 or lower on gonioscopy examination), history of angle-closure glaucoma, or previous iridotomy |
| 4.05 | History of iris trauma, Adie's tonic pupil, abnormal pupil shape in either eye, or anisocoria > 1 mm between pupils under mesopic conditions at the screening visit |
| 4.06 | Lens opacity in either eye that is determined to cause significant disturbance of the central visual axis on screening biomicroscopy |
| 4.07 | Diagnosis of any type of glaucoma or ocular hypertension |
| 4.08 | Bifocal or multifocal spectacles or contact lenses for habitual correction. Participants willing to wear study-provided monofocal correction (either spectacles or contact lenses) during the study can be enrolled |
| 4.09 | Abnormal and clinically significant results according to the investigator or designee, on physical/ophthalmic examination or medical history |



| 5. | Other |
|---|---|
| 5.01 | Females who are pregnant, nursing, or planning a pregnancy during the study. |



#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAE.

Individuals who do not meet the criteria for participation in this study (screen failures) may not be rescreened.



# 6. Study Intervention

Study intervention is defined as any investigational intervention intended to be administered to a study participant according to the study protocol.

6.1. Study Intervention(s) Administered

| <b>Study Intervention Name</b> | AGN-190584 | Vehicle |
|---|---|---|
| Dosage Formulation | Topical eye drop | Topical eye drop |
| Identity of Formulation | Pilocarpine HCl 1.25% Ophthalmic Solution | Pilocarpine HCl Placebo Ophthalmic<br>Solution |
| · | | |
| Drug Substance | Pilocarpine 1.25% | Not applicable |
| Route of Administration | Topical eye drop | Topical eye drop |
| <b>Dosing Instructions</b> | 1 drop in each eye once daily | 1 drop in each eye once daily |
| Manufacturer Number and Timing of | Allergan Sales, LLC. | Allergan Sales, LLC. |

As this is a double-masked study, AGN-190584 and Vehicle will be supplied in identically appearing bottles and cartons.









# 6.2. Preparation/Handling/Storage/Accountability

The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.



Only participants enrolled in the study may receive study intervention, and only authorized site staff may supply or administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff. All study intervention must be stored upright, in a refrigerator, and protected from freezing.

Participants will be instructed on the proper storage of study intervention and to keep it out of the reach of children at all times.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

All participants will be centrally assigned to randomized study intervention using the IxRS. Randomization and kit assignment will be conducted on Day 1 (baseline). At Day 1, participants will be randomized in a 1:1 ratio into 1 of the 2 study groups. This randomization will be stratified by age (2 groups:  $\leq 50$  years and > 50 years), baseline binocular DCNVA (2 groups: 20/40 to 20/60 inclusively, and worse than 20/60), iris color (brown and non-brown), and emmetropes/non-emmetropes. A maximum of 50% (75 per arm) of the participants enrolled will have brown iris color, and a maximum of 25% (38 per arm) of the participants will be non-emmetropes (a sphere outside of -0.50 D to +0.75 D and/or a cylinder greater than 0.75 D).







## **6.5.** Concomitant Therapy

The use of any concomitant medication, prescription or over-the-counter, is to be recorded on the participant's eCRF at each visit along with the reason the medication is taken.

From screening to the EOS, site staff will question each participant specifically on the use of concomitant medications. Site staff must notify the sponsor immediately if a participant consumes any concomitant medications not permitted by the protocol. Participants who used prohibited concomitant medications may be discontinued from the study at the discretion of the investigator or the sponsor.

#### 6.5.1. Prohibited Interventions and Washout Before the Study

Use of medications that may have a substantial effect on visual function or the optical properties of the eye is prohibited 2 weeks prior to Day 1 visit and during the study:

- systemic medications with potential ocular side effects, including topiramate, hydroxychloroquine, ethambutol, phosphodiesterase 5 inhibitors (sildenafil, vardenafil, tadalafil), or tamoxifen
- ophthalmic, systemic, or intranasal anticholinergics and α-adrenergic receptor agonists with potential pupillary or accommodative effects, including oxymetazoline, pilocarpine, tetrahydrozoline, phenylephrine, naphazoline, cyclopentolate, atropine, beta-blockers, or antihistamines
- systemic maprotiline, tricyclic antidepressants, or monoamine oxidase inhibitors



#### **6.5.2.** Permitted Interventions

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the participant is receiving at the time of enrollment or receives during the study must be recorded along with:

- Indication
- Dates of administration including start and end dates
- Dosage information including dose and frequency

Therapy considered necessary for the participant's welfare may be given at the discretion of the investigator. If the permissibility of a specific medication/intervention is in question, please contact the sponsor.

The sponsor or designee should be contacted if there are any questions regarding concomitant or prior therapy.

The concurrent use of nonocular medications that do not have a substantial effect on the pupil, accommodative properties, or retinal function of the eye will be permitted during the study if a stable dosing regimen is established. The dosing regimen is not considered to be stable if a participant starts, stops, or changes the dose/drug during the study.

Any medication taken during the study between the date of the first dose of study intervention and the date of the EOS visit will be recorded in the eCRF as a concomitant medication; any medication started after the EOS visit will not be considered a concomitant medication and should not be captured in the eCRF.

#### 6.5.3. Rescue Medicine

Rescue medicine is not applicable.

#### 6.5.4. Prohibited Interventions During the Study

Use of ocular medications other than study intervention or medications administered to conduct study procedures are prohibited from the screening visit until study exit.

The decision to administer a prohibited medication/treatment will be made with the safety of the study participant as the primary consideration. When possible, Allergan should be notified before the prohibited medication/treatment is administered.

#### 6.6. Dose Modification

Dose modification is not applicable.

## 6.7. Intervention after the End of the Study

No interventions after the end of the study are planned.



# 7. Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

A premature discontinuation will occur if a participant who signs the ICF and is dosed ceases participation in the study, regardless of circumstances, before the completion of the protocol-defined study procedures.

Reasons for discontinuation from the study intervention and/or the study may include the following:

- AE
- Lack of efficacy
- Lost to follow-up
- Noncompliance with study drug
- Physician decision
- Pregnancy
- Protocol deviation
- Site terminated by sponsor
- Study terminated by sponsor
- Withdrawal by subject
- Death
- Other

# 7.1. Discontinuation of Study Intervention

See the SoA (Section 1.3) for data to be collected at the time of early exit.

Participants who discontinue the study intervention early will be encouraged to stay in the study for the safety assessments at Day 30.

# 7.2. Participant Discontinuation/Withdrawal from the Study

 A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.



- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.
- See the SoA (Section 1.3) for data to be collected at the time of early exit.

# 7.3. Lost to Follow Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts will be documented in the participant's medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.



#### 8. Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA (Section 1.3). Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor promptly upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria. The investigator will maintain a screening log to
  record details of all participants screened and to confirm eligibility or record reasons for
  screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (eg, blood count) and obtained before signing of the ICF may be utilized for screening or baseline purposes provided the procedures met the protocol-specified criteria and were performed within the timeframe defined in the SoA.
- The maximum amount of blood collected for PK from each participant over the duration
  of the study, including any extra assessments that may be required, will not exceed 45 mL.
  Repeat or unscheduled samples may be taken for safety reasons or for technical issues
  with the samples.

# 8.1. Efficacy Assessments

Efficacy assessments are: mesopic and photopic, high contrast DCNVA for each eye and binocularly, mesopic and photopic, high contrast DCIVA for each eye and binocularly, PRO questionnaires (NVPTQ, PICQ,



**Table 8-1 Efficacy Assessments** 

| Assessment | Timing | Measurement |
|---|---|---|
| Visual Acuity | | |
| Mesopic, high contrast<br>DCNVA for each eye and<br>binocularly | <ul> <li>Screening</li> <li>Days 1, 14, and 30: Hours 0, 0.25, 0.5, 1, 3, 6, 8, and 10</li> <li>Days 3 and 7: Hours 0, 1, and 3</li> </ul> | <ul> <li>Visual acuity for near (40-cm), intermediate (66-cm) and distance (4-meter) targets will be measured in mesopic and photopic conditions.</li> <li>Mesopic condition is defined as lighting 3.2 to 3.5 candelas per square meter (cd/m²; 10 to 11 lux) measured at the target.</li> <li>Photopic condition is defined as lighting ≥ 80 cd/m² (251 lux) measured at the target.</li> </ul> |
| Photopic, high contrast<br>DCNVA for each eye and<br>binocularly | <ul> <li>Screening</li> <li>Days 1, 14, and 30: Hours 0, 0.25, 0.5, 1, 3, 6, 8, and 10</li> <li>Days 3 and 7: Hours 0, 1, and 3</li> </ul> | |
| Mesopic and photopic,<br>high contrast DCIVA for<br>each eye and binocularly | <ul> <li>Screening</li> <li>Days 1, 14, and 30: Hours 0, 1, 3, 6, 8, and 10</li> <li>Days 3 and 7: Hours 0, 1, and 3</li> </ul> | |





| Assessment | Timing | Measurement |
|---|---|---|
| PRO Questionnaires | | |
| Mesopic and Photopic<br>NVPTQ | <ul><li>Day 1, Hour 0</li><li>Day 14, Hour 1</li><li>Day 30, Hour 3</li></ul> | <ul> <li>Comprised of 12 questions on 4 reading tasks (ie, reading a paragraph from a book, reading excerpts from an article in a newspaper, reading a portion of a nutrition label, and reading a section from a restaurant menu)</li> </ul> |
| | | <ul> <li>Participants will complete specific reading tasks<br/>under mesopic and photopic conditions without<br/>any near-vision correction</li> </ul> |
| | | <ul> <li>Participants will then answer 3 questions for each<br/>task, rating their vision-related reading ability and<br/>satisfaction with their vision-related reading<br/>ability</li> </ul> |
| | | <ul> <li>There is no explicit recall period used for the<br/>NVPTQ; the intention is for patients to complete<br/>the NVPTQ immediately after completing each<br/>task.</li> </ul> |
| | | <ul> <li>For more details on instructions and questions in<br/>NVPTQ, please see Appendix 8</li> </ul> |
| PICQ | <ul><li>Day 1, Hour 0</li><li>Day 30, Hour 3</li></ul> | <ul> <li>Participants will answer 20 questions about the<br/>degree to which they were impacted by their<br/>difficulty seeing up close (eg, found daily near-<br/>vision tasks difficult, or experienced self-<br/>consciousness); or engaged in coping behaviors<br/>(eg, changed the font size on electronic screens)<br/>during the previous 7 days</li> </ul> |
| | | <ul> <li>For more details on instructions and questions in<br/>PICQ, please see Appendix 8</li> </ul> |




### 8.2. Safety Assessments

Planned timepoints for all safety assessments are provided in the SoA (Section 1.3).

#### 8.2.1. Vital Signs

Vital signs will be assessed as follows:

- Blood pressure and pulse rate will be assessed.
- Systolic and diastolic blood pressure will be measured using an appropriate sphygmomanometer after participants have been at rest (seated) for at least 5 minutes. Blood pressure will be recorded in mm Hg.
- Heart rate will be measured in bpm after the participant has been in a resting state (seated) for at least 5 minutes. Pulse will be counted for 30 seconds, multiplied by 2, and recorded in bpm.
- Blood pressure and pulse measurements will be assessed with a completely automated device. Manual techniques will be used only if an automated device is not available.
   Manual techniques will be used only by adequately trained personnel; whenever possible, the same person should perform all manual assessments as much as possible.
- Participants should refrain from smoking or ingesting caffeine during the 30 minutes preceding the measurement.

#### 8.2.2. Pregnancy Testing

Pregnancy test kits will be provided by the investigator and will be administered according to the instructions provided with the tests. WOCBP must have a negative test result before receiving



study intervention. This test will also be performed at the Day 30 (Early Exit) visit, and may be performed at any other visit, at the investigator's discretion. At each visit, the investigator should discuss contraceptive use compliance with WOCBP. Additional details are provided in Appendix 6.

# 8.2.3. Photopic and Mesopic, High Contrast Corrected Distance Visual Acuity for Each Eye and Binocularly

Photopic and mesopic, high contrast CDVA, for each eye and binocularly, will be assessed using the provided visual acuity charts for distance vision in a room with mesopic lighting conditions (defined by lighting 3.2 to 3.5 candelas  $[cd]/m^2$  [10 to 11 lux] measured at the target) and photopic lighting conditions (defined by lighting  $\geq 80$  cd/m<sup>2</sup> [251 lux] measured at the target). Forced choice letter by-letter scoring will be used for each test and the total number of correct letters or the highest value (number) of the grid identified (as applicable) will be recorded. Further details are outlined in the Procedure Manual.

#### 8.2.4. Near Contrast Sensitivity

Near contrast sensitivity assessment will be conducted under photopic conditions. A Pelli-Robson contrast sensitivity chart will be used. The logarithmic contrast sensitivity value of the last triplet of which at least 2 letters are correctly read is marked as the contrast sensitivity. Further details are outlined in the Procedure Manual.

#### 8.2.5. Study Intervention Tolerability and Drop Comfort Assessments

The presence and severity of ocular symptoms will be elicited from the participant for both eyes after dosing. Symptoms, including blurred vision, foreign body sensation, pain, burning/stinging, tearing, and itching, will be classified using a 5-point grading scale with 0 = none, +0.5 = trace, +1 = mild, +2 = moderate, and +3 = severe. The duration of symptoms (< 1 minute, 1 to 5 minutes, > 5 minutes) will be captured once immediately after the second eye is instilled with a drop of study intervention. If any other ocular symptoms are present, these will also be captured.

Participants will be asked to rate the overall comfort of the eye drops using a 6-point scale (ie, soothing, very comfortable, comfortable, uncomfortable, very uncomfortable, and intolerable) immediately after the second eye is instilled with a drop of study intervention, for both eyes.

#### 8.2.6. Temporal/Supraorbital Headache Visual Analog Scale

Participants will be asked to rate the degree of temporal and supraorbital headache experienced after the second eye is instilled with a drop of study intervention, for the right and left eyes separately. Headache will be reported on an unmarked 100-mm wide VAS, ranging from no pain on the left to worst possible pain on the right.



#### 8.2.7. Intraocular Pressure

IOP must be measured after the biomicroscopic exam is completed and prior to pupil dilation. Measurements will be taken using a Goldmann applanation tonometer affixed to a slit-lamp with the participant seated. The participant and slit-lamp should be adjusted so that the participant's head is firmly positioned on the chin rest and against the forehead rest without leaning forward or straining. Tight fitting neckwear should be loosened. Both eyes will be tested, with the right eye preceding the left eye. The measurer will look through the binocular viewer of the slit lamp at low power. The tension knob will be preset at a low-pressure value (4 to 6 mm Hg). The measurer will follow the image of the fluorescein stained semicircles while slowly rotating the tension knob until the inner borders of the fluorescein rings touch each other at the midpoint of their pulsation in response to the cardiac cycle. When this image is reached, the measurer will take his/her fingers off the tension knob and record the IOP reading along with the date and time of day.

#### 8.2.8. Slit-lamp Biomicroscopy

Biomicroscopic examinations will be performed using a slit-lamp. The examinations will include evaluation of the condition of the eyelids, conjunctiva, cornea, anterior chamber, and iris/pupil.



# **Eyelid/Eyelid Margins/Lashes:**

| Fd | em | เฉ |
|----|-----|----|
| EU | CII | la |

| 0 | (None) | = | No edema |
|---|---|---|---|
| +0.5 | (Trace) | = | Localized, minimal (trace) swelling |
| +1 | (Mild) | = | Localized, mild swelling |
| +2 | (Moderate) | = | Diffuse, moderate swelling |
| +3 | (Severe) | = | Diffuse, severe swelling |
| <b>Erythema</b> | | | |
| 0 | (None) | = | No erythema |
| +0.5 | (Trace) | = | Localized, minimal (trace) flush reddish color |
| +1 | (Mild) | = | Localized, mild, flush reddish color |
| +2 | (Moderate) | = | Diffuse reddish color encompassing the entire lid margin |
| +3 | (Severe) | = | Deep diffuse reddish color of lid margins and superior |

# Conjunctiva (Bulbar):

## **Hyperemia**

| 0 | (None) | = | No hyperemia |
|--------------|------------|---|--------------------------------------|
| +0.5 | (Trace) | = | Minimal (trace) flush, reddish color |
| +1 | (Mild) | = | Mild flush, reddish color |
| +2 | (Moderate) | = | Bright red color |
| +3 | (Severe) | = | Deep, bright diffuse redness |
| <u>Edema</u> | | | |
| 0 | (None) | = | No edema |
| +0.5 | (Trace) | = | Localized, minimal (trace) swelling |
| +1 | (Mild) | = | Localized, mild swelling |
| +2 | (Moderate) | = | Diffuse, moderate swelling |
| +3 | (Severe) | = | Diffuse, severe swelling |



## Conjunctiva (Palpebral):

# **Hyperemia**

| 0 | (None) | = | No hyperemia |
|--------------|------------|---|--------------------------------------|
| +0.5 | (Trace) | = | Minimal (trace) flush, reddish color |
| +1 | (Mild) | = | Mild flush, reddish color |
| +2 | (Moderate) | = | Bright red color |
| +3 | (Severe) | = | Deep, bright diffuse redness |
| <u>Edema</u> | | | |
| 0 | (None) | = | No edema |
| +0.5 | (Trace) | = | Localized, minimal (trace) swelling |
| +1 | (Mild) | = | Localized mild swelling |

# +1 (Mild) = Localized, mild swelling

+2 (Moderate) = Diffuse, moderate swelling +3 (Severe) = Diffuse, severe swelling

#### Cornea:

#### Edema

| 0 | (None) | = | No edema |
|---|---|---|---|
| +0.5 | (Trace) | = | Localized, minimal (trace) epithelial haze |
| +1 | (Mild) | = | Dull glass appearance of epithelium that may include fine localized microcystic changes |
| +2 | (Moderate) | = | Dull glass appearance of the epithelium with large<br>number of cystic changes with or without stromal edema |
| +3 | (Severe) | = | Epithelial bullae and/or stromal edema, localized or diffuse, with or without stromal striae |

## Superficial Punctate Keratopathy

| ( | ) = | No su | perficial | punctate | keratopath | y |
|---|-----|-------|-----------|----------|------------|---|
|---|-----|-------|-----------|----------|------------|---|

+0.5 = Trace +1 = Mild +2 = Moderate +3 = Severe

#### **Anterior Chamber:**

The anterior chamber will be evaluated for pathology. If pathology is present, it will be described.



#### Iris/Pupil:

The iris/pupil will be evaluated for pathology. If pathology is present, it will be described.

#### 8.2.9. Manifest Refraction

Manifest refraction (distance and near) will be performed according to standard clinical practice in both mesopic and photopic conditions.

If a participant loses  $\geq 1$  line of CDVA or DCNVA compared with Hour 0 of the same study visit at Hour 1 after dosing, a manifest refraction should be repeated under the same lighting conditions.

Additional details are outlined in the Procedure Manual.

#### **8.2.10.** Dilated Funduscopic Examination

The fundus assessments should be conducted through a dilated pupil. The examinations will include evaluation of the lens, vitreous, fundus, and optic nerve. The C/D ratio will be assessed. The investigator should note if the pupil dilated normally.

#### Lens:

#### Lens Assessment:

Use biomicroscopic examination, indirect lenses, direct/indirect ophthalmoscopy, etc., as appropriate, to visualize.

#### Lens Status:

The lens will be evaluated for pathology. If pathology is present, it will be described.

#### Cataract Assessment:

Under dilated examination, the presence and severity of nuclear, cortical, and posterior subcapsular cataract lens opacities will be evaluated. At the first dilated examination, each type of cataract, if present, will be graded using the scale below. At the last follow-up dilated examination, each type of cataract will be assessed for change from baseline and if changed, the current severity will be graded using the scale below:

0 = None

+1 = Mild

+2 = Moderate

+3 = Severe

#### **Vitreous:**

The vitreous will be evaluated for pathology. If pathology is present, it will be described. It will be noted if the condition is not evaluable.



#### **Fundus:**

The fundus (posterior pole; periphery, when dilated) will be evaluated for pathology. If pathology is present, it will be described. It will be noted if the condition is not evaluable.

#### **Optic Nerve:**

The optic nerve will be evaluated for pathology. If pathology is present, it will be described. It will be noted if the condition is not evaluable.

#### C/D Ratio:

C/D ratio will be reported using a 0.0 to 1.0 scale. It will be noted if the condition is not evaluable.

#### 8.2.11. Suicidal Risk Monitoring

Suicidal risk monitoring is not applicable to this ophthalmology study.

#### 8.3. Adverse Events and Serious Adverse Events

The definitions of an AE or SAE can be found in Appendix 2.

AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study intervention (ie, repeat treatment) or study (see Section 7).

# 8.3.1. Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

All SAEs from the signing of the ICF until 30 days after the last dose of study intervention will be collected at the timepoints specified in the SoA (Section 1.3), and as observed or reported spontaneously by study participants.

All AEs from the signing of the ICF until 30 days after the last dose of study intervention will be collected at the timepoints specified in the SoA (Section 1.3), and as observed or reported spontaneously by study participants.

Medical occurrences that begin before the start of study intervention, but after obtaining informed consent will be recorded in the AE section of the eCRF.

All SAEs will be recorded and reported to the sponsor or designee within 24 hours, as indicated in Appendix 2. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.



Investigators are not obligated to actively seek AE or SAE information after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

The methods of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 2.

#### 8.3.2. Method of Detecting Adverse Events and Serious Adverse Events

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

#### 8.3.3. Follow-up of Adverse Events and Serious Adverse Events

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All AEs/SAEs will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3).

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by Allergan to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

If a participant dies during participation in the study, the investigator will provide Allergan with a copy of any postmortem findings including histopathology.

If a participant is hospitalized and discharged, follow-up attempts must be made to obtain the discharge summary from the hospital and, if obtained, it should be sent to the sponsor.

New or updated information will be recorded in the originally completed eCRF.

The investigator will submit any updated SAE data to Allergan within 24 hours of receipt of the information.

#### 8.3.4. Regulatory Reporting Requirements for Serious Adverse Events

- Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/IECs, and investigators.



- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing an SAE or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

#### 8.3.5. Pregnancy

- If a pregnancy is confirmed after the participant has received the study intervention, the participant may choose to exit the study after appropriate safety follow-up or to remain in the study for all safety and efficacy follow-up assessments through the EOS visit.
- Details of all pregnancies in female participants and, if indicated, female partners of male participants will be collected after the start of study intervention and through the duration of the pregnancy.
- If a pregnancy is reported, the investigator should inform Allergan within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 6.
- Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) or genetic abnormalities (whether leading to an elective abortion or not) are considered SAEs.

#### **8.3.6.** Medication Errors

Medication error refers to any unintended error in the dosing and/or administration of the study intervention as per instructions in the protocol. Medication errors generally fall into 4 categories as follows:

- Wrong study drug
- Wrong dose (including dosing regimen, strength, form, concentration, amount)
- Wrong route of administration
- Wrong participant (ie, not administered to the intended participant)

#### 8.4. Treatment of Overdose

Treatment of overdose is not applicable to this ophthalmology study.



#### 8.5. Pharmacokinetics

Blood samples for quantitation of pilocarpine in participant's plasma will be collected from approximately 10% of enrolled participants at selected sites.

#### 8.5.1. Blood Pharmacokinetic Sampling Procedure

- A qualified phlebotomist will collect 5 mL of each participant's blood via an indwelling catheter or venipuncture from either arm into one 6 mL vacutainer tube containing K<sub>2</sub>EDTA as an anticoagulant.
- Plasma samples of approximately 2.5 mL will be separated from each blood sample collected for measurement of plasma concentrations of pilocarpine as specified in the SoA (Section 1.3).
- Instructions for the collection and handling of biological samples will be provided by Allergan. The actual date and time (24-hour clock time) of each sample will be recorded. PK blood samples to determine pilocarpine concentrations should be drawn at the nominal times, relative to the dosing time, and the actual time of the blood draw must be recorded in the source documents and eCRFs. Samples taken outside the allowable time window will be noted as protocol deviations, and the reason for deviation must be recorded in the source documents and eCRFs. Predose samples must be drawn within 15 minutes of the dosing time.
- Study center staff will record the atomic clock times of all blood draws for each
  participant and will label vacutainer and polypropylene tubes with a coded label that
  corresponds to the participant number and blood draw time. The central lab will supply
  the coded labels, vacutainers, and polypropylene tubes. The study center will be
  responsible for all other supplies.
- Samples will be used to evaluate the pharmacokinetics of pilocarpine. Each plasma sample will be divided into 2 aliquots (1 each for primary and backup PK samples). Samples collected for analyses of pilocarpine plasma concentration may also be used to evaluate safety or efficacy aspects related to concerns arising during or after the study.

Drug concentration information that would unmask the study will not be reported to investigative sites or blinded personnel until the study has been unmasked.

Bioanalytical representatives will be unmasked for PK sample bioanalysis during the conduct of the study. The unmasking of bioanalytical representatives is to be carried out in a secure manner following Allergan's standard operating procedures. Extreme care and diligence will be taken to ensure no other individuals outside the bioanalytical team will be unblinded.



#### **Blood Volume Collected per Participant**

- Approximately 10% of participants at selected sites
- PK blood samples: 45 mL (9 blood samples, 5 mL each)

Within 30 minutes from the time of the blood draw, blood samples must be centrifuged at no less than 2000 g for 15 minutes at approximately  $4^{\circ}$ C. After centrifugation, the plasma samples will be harvested and aliquoted into two approximately 1.25 mL samples in cryovials (one primary and one backup). The samples should be placed on wet ice immediately after aliquoting and transferred to a  $-20^{\circ}$ C freezer within one hour of processing to plasma.

Study center staff will send plasma samples to the central lab for storage at the end of each period. Before shipment and on the day of shipment, the sponsor and the central lab will be notified by email as to the time and method of shipment. Primary and backup samples will be shipped to the central lab in separate shipments on separate days.

#### 8.5.2. Pharmacokinetic Sample Bioanalysis

Plasma concentrations of pilocarpine in plasma will be determined using validated liquid chromatography-tandem mass spectrometry methods.

### 8.6. Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

#### 8.7. Genetics

Genetics are not evaluated in this study.

#### 8.8. Biomarkers and Other Assessments

#### 8.8.1. Biomarkers

Biomarkers are not evaluated in this study.

#### **8.8.2.** Determination of Dominant Eye

Participants will be asked to extend their arms out in front of them at eye level, with their palms facing away, fingers together, and facing upward. Participants will bring their hands together, forming a small window by overlapping their thumbs and overlapping their fingers. Participants will select a small object at least 10 feet in front of them and look at it with both eyes through the view window in their hands. While remaining focused on the object, participants will close the right eye and take note of whether the image remains visible. If the image remains visible, the left eye is the dominant eye. If the image is no longer visible, the right eye is the dominant eye. This will be confirmed by closing the left eye and taking note of whether the image remains visible. Details will be outlined in the Procedure Manual.



### 8.9. Health Economics

PRO instruments (questionnaires) are administered in this study

At screening, participants will answer questions on vision functioning and health-related quality of life using the NEI VFQ-25, including the near vision subscale items (Questions A3 to A5) from the Appendix of Optional Additional Questions.

Each participant will also perform four different near vision reading tasks under mesopic and photopic conditions. Participants will subsequently rate their vision-related reading ability, and satisfaction with their vision-related reading ability on the NVPTQ.

Participants will also answer questions measuring overall satisfaction with the treatment using questions assessing the impact of presbyopia on their life – and need for compensatory coping mechanisms – using the PICQ.

#### 9. Statistical Considerations

# 9.1. Statistical Hypotheses

The null and alternative hypotheses for the primary efficacy endpoint are:

- H<sub>0</sub>: AGN-190584 ophthalmic solution and vehicle dosed bilaterally, once daily for 30 days have the same effect in the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 3;
- H<sub>A</sub>: AGN-190584 ophthalmic solution and vehicle dosed bilaterally, once daily for 30 days do not have the same effect in the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 3.

The null and alternative hypotheses for the key secondary efficacy endpoint are:

• H<sub>0</sub>: AGN-190584 ophthalmic solution and vehicle dosed bilaterally, once daily for 30 days have the same effect in the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 6;



• H<sub>A</sub>: AGN-190584 ophthalmic solution and vehicle dosed bilaterally, once daily for 30 days do not have the same effect in the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 6.

## 9.2. Sample Size Determination

The primary efficacy endpoint is the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 3. The key secondary efficacy endpoint is the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 6. The sample size calculation is based on the key secondary efficacy endpoint. The vehicle group intervention effect is assumed to be 3.6%, as observed in the Phase 2 study. AGN-190584 effect is assumed to be 16% in emmetropes and 12% in non-emmetropes. This gives an overall AGN-190584 effect of 15% assuming emmetropes will be 75% of the study population. 135 participants will be required in each study intervention group to detect the above difference with a power of 90% or greater at the 2-sided 5% significance level. Assuming a 10% dropout rate, approximately 150 participants per study intervention group will be randomized.

## 9.3. Populations for Analyses

The analysis populations will consist of participants as defined below:

- The ITT population includes all randomized participants. Participants will be summarized according to the randomized study intervention.
- The safety population includes all treated participants who receive ≥ 1 administration of study intervention. Participants will be summarized according to the study intervention they actually received.

# 9.4. Statistical Analyses

The SAP will be developed and finalized before database lock and unmasking and will describe the participant populations to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary and secondary endpoints.

#### 9.4.1. Efficacy Analyses

The efficacy analyses will be based on the ITT population. Baseline for efficacy is defined as the last nonmissing efficacy assessment before the first dose of study intervention. All statistical tests will be 2-sided hypothesis tests performed at the 5% level of significance for main effects. All confidence intervals will be 2-sided 95% confidence intervals, unless stated otherwise.



#### 9.4.1.1. Analysis Endpoints

The primary and secondary efficacy endpoints are listed below and analyses will be described in the following sections. The analyses for other efficacy endpoints listed below will be described in the SAP.

#### **Primary Efficacy Endpoint:**

 Proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 3.

#### **Key Secondary Efficacy Endpoint:**

• Proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 6.

#### **Secondary Efficacy Endpoints:**

- 1. Proportion of participants gaining 3-lines or more in mesopic, high contrast, binocular, DCNVA at Day 30, Hour 8.
- 2. Change from baseline mesopic, high contrast, binocular DCNVA letters at Day 30, Hour 0.5.
- 3. Proportion of participants achieving 20/40 or better in photopic, high contrast, binocular, DCNVA at Day 30, Hour 1.
- 4. Mesopic NVPTQ Performance score mean change from baseline at Day 30, Hour 3.
- 5. Change from baseline photopic, high contrast, binocular DCIVA letters at Day 30, Hour 3.
- 6. Proportion of participants gaining 3-lines or more in mesopic, high contrast, binocular, DCNVA at Day 30, Hour 10.
- 7. Change from baseline mesopic, high contrast, binocular DCNVA letters at Day 30, Hour 0.25.
- 8. Proportion of participants achieving 20/40 or better in photopic, high contrast, binocular, DCNVA at Day 30, Hour 3.
- 9. Mesopic NVPTQ Satisfaction score mean change from baseline at Day 30, Hour 3.
- 10. PICQ Coping score mean change from baseline at Day 30, Hour 3.
- 11. PICQ Impact score mean change from baseline at Day 30, Hour 3.



#### 9.4.1.2. Primary Analyses

The proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 3 will be analyzed using chi-square test. Missing data will be regarded as 3-line gain failure.

#### 9.4.1.3. Secondary Analyses

The key secondary efficacy endpoint is the proportion of participants gaining 3 lines or more in mesopic, high contrast, binocular DCNVA at Day 30, Hour 6.

The key secondary efficacy endpoint will be analyzed using a chi-square test. Missing data will be regarded as 3-line gain failure.

All analyses for other secondary efficacy endpoints will be based on observed data only. Secondary endpoints 1, 3, 6, and 8 will be analyzed using a chi-square test. Secondary endpoints 2, 4, 5, and 7 will be analyzed using MMRM with study intervention group, visit, visit by study intervention group interaction, age group, baseline binocular DCNVA severity, iris color, emmetropes/non-emmetropes, baseline value, and baseline value by visit interaction as fixed effects. The within-participant correlation error structure is unstructured. Secondary endpoints 9, 10, and 11 will be analyzed using analysis of covariance with study intervention group, age group, baseline binocular DCNVA severity, iris color, emmetropes/non-emmetropes, and baseline domain score as fixed effects.

To control the overall Type 1 error rate in the efficacy analysis, a sequential testing procedure will be used. The test for the key secondary endpoint will be implemented only if the primary efficacy endpoint yields statistically significant results. All other secondary efficacy endpoints will be tested only if the key secondary efficacy endpoint is statistically significant. A proper multiple comparison procedure will be pre-specified in the SAP.

#### 9.4.2. Safety Analyses

The safety analysis will be performed using the safety population and will be fully defined in the SAP. The safety parameters will include AEs, vital signs (blood pressure and heart rate), mesopic and photopic, high contrast, binocular CDVA, near contrast sensitivity, study intervention tolerability and drop comfort assessments, temporal/supraorbital headache assessment using VAS, IOP, slit-lamp biomicroscopy, manifest refraction, dilated funduscopic examination, and pregnancy test. For each safety parameter, the last nonmissing safety assessment before the first dose of study intervention will be used as the baseline.



#### 9.4.2.1. Adverse Events

An AE will be considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date of the first dose of study intervention. However, an AE that occurs more than 30 days after the last dose of study intervention will not be counted as a TEAE.

An AE will be considered a treatment-emergent SAE if it is a TEAE that additionally meets any SAE criteria.

The number and percentage of participants reporting TEAEs during the study will be tabulated by system organ class and preferred term and by system organ class, preferred term, and severity.

If more than one AE is coded to the same preferred term for the same participant, the participant will be counted only once for that preferred term using the most severe and most related occurrence for the summarizations by severity and by relationship to study intervention.

Summary tables will be provided for participants with SAEs and participants with AEs leading to discontinuation if 5 or more participants reported such events. Listings of all AEs, SAEs, and AEs leading to discontinuation by participant will be presented.

#### 9.4.2.2. Other Safety Analyses

All other safety variables will be analyzed with descriptive statistics. Detailed methods for the analysis of other safety variables will be described in the SAP.

#### 9.4.3. Pharmacokinetic Analyses

#### 9.4.3.1. Pharmacokinetic Parameters

The following PK parameters will be calculated based on standard Phoenix WinNonlin equations:  $AUC_{0-last.ss}$ , maximum plasma drug concentration at steady state, time of maximum plasma drug concentration at steady state,  $C_{min,ss}$ , and peak-to-trough ratio.

 $C_{min,ss}$  will be determined observationally as the drug concentration during the dosing interval at steady state.

AUC<sub>0-last,ss</sub> will be calculated by using the linear-log trapezoidal rule.

#### 9.4.3.2. Statistical Analyses of Pharmacokinetic Data

Details of the statistical analyses of PK data will be described in the pharmacokinetic analysis plan finalized before database lock.



# 9.5. Interim Analyses

No interim analysis is planned.

# 9.5.1. Data Monitoring Committee

Not applicable.



# 10. Supporting Documentation and Operational Considerations



# 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

#### 10.1.1. Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines
  - o Applicable ICH/International Organization for Standardization GCP guidelines
  - o Applicable laws and regulations
- The protocol, protocol amendments, ICF, IB, and other relevant documents (eg, advertisements) must be submitted to an IRB/IEC by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
  - o Providing oversight of the overall conduct of the study at the site and adherence to requirements of applicable local regulations, for example 21 CFR, ICH guidelines, the IRB/IEC, and European regulation 536/2014 for clinical studies (if applicable)





#### 10.1.3. Informed Consent Process

- The investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, Health Insurance Portability and Accountability Act requirements, where applicable, and the IRB/IEC or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.

#### 10.1.4. Data Protection

- Participants will be assigned a unique identifier. Any participant records or datasets that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection laws. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

#### 10.1.5. Posting Clinical Study Data

- Study data and information may be published in nonpromotional, peer-reviewed publications either by or on behalf of the sponsor.
- Clinical study reports, safety updates, and annual reports will be provided to regulatory authorities as required.
- Company-sponsored study information and tabular study results will be posted on the United States National Institutes of Health's website www.ClinicalTrials.gov and other publicly accessible sites



#### **10.1.6.** Data Quality Assurance

- All participant data relating to the study will be recorded on printed or electronic CRFs unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.
- Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICFs, pertaining to the conduct of this study must be retained by the investigator as stated in the clinical trial agreement. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### **10.1.7.** Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data reported on the CRF or entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study.
- Definition of what constitutes source data can be found in Section 4.0 of ICH E6, GCP: Consolidated Guidance and records must be attributable, legible, contemporaneous, original, and accurate.







#### 10.1.9. Publication Policy

- Allergan as the sponsor has proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple investigators and sites and Allergan personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.
- The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

#### 10.1.10. Compliance with Protocol

The investigator is responsible for compliance with the protocol at the investigational site. A representative of the sponsor will make frequent contact with the investigator and his/her research staff and will conduct regular monitoring visits at the site to review participant and study intervention accountability records for compliance with the protocol. Protocol deviations will be discussed with the investigator upon identification. The use of the data collected for the participant will be discussed to determine if the data are to be included in the analysis. The investigator will enter data that may be excluded from analysis as defined by the protocol deviation specifications. Significant protocol deviations will be reported to the IRB/IEC according to the IRB/IEC's reporting requirements.



# 10.2. Appendix 2: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definition of AE**

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### **AESI**

An AESI (serious or nonserious) is one of scientific and medical concern specific to the sponsor's study drug/device or program, which warrants ongoing monitoring and rapid communication by the investigator to the sponsor. Such an event might warrant further investigation in order to characterize and understand it.

There are no AESIs identified for the study intervention AGN-190584.

#### **Events Meeting the AE Definition**

- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition
- New condition detected or diagnosed after study intervention administration even though it may have been present before the start of the study
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction
- Lack of efficacy or failure of expected pharmacological action per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from the lack of efficacy will be reported as AEs or SAEs if they fulfill the definition of an AE or SAE.



#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease or disease progression, unless judged by the investigator to be more severe than expected for the participant's condition. Merely repeating an abnormal test, in the absence of any of the above conditions. Any abnormal test result that is determined to be an error does not require recording as an AE.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital)
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen

#### **Definition of SAE**

SAEs must meet both the AE criteria described above and the seriousness criteria listed below.

#### An SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

#### b. Is life threatening

The term *life threatening* in the definition of *serious* refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or intervention that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether hospitalization occurred or was necessary, the AE should be considered serious.

Hospitalization for elective intervention of a pre-existing condition that did not worsen from baseline is not considered an AE.



### d. Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other situations:

Medical or scientific judgment should be exercised in deciding whether SAE
reporting is appropriate in other situations such as important medical events that may
not be immediately life threatening or result in death or hospitalization but may
jeopardize the participant or may require medical or surgical intervention to prevent
one of the other outcomes listed in the above definition. These events should usually
be considered serious.

Examples of such events include invasive or malignant cancers, intensive intervention in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

#### Recording and Follow-Up of AEs and/or SAEs

#### **AE and SAE Recording**

- When an AE or SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE or SAE information in the eCRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Allergan in lieu of completion of the AE or SAE eCRF page.
- There may be instances when copies of medical records for certain cases are requested by Allergan. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Allergan.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.



| Assessment of | Assessment of Intensity |
|---|---|
| MILD | A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. |
| MODERATE | A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. |
| SEVERE | A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. |

An event is defined as *serious* when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE.
- A *reasonable possibility* of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to Allergan. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to Allergan.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality



#### assessment.

• The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### **Reporting of SAEs**

#### **SAE/SADE** Reporting

- Email is the preferred method to transmit SAE information. The email address is IR-Clinical-SAE@allergan.com.
- Facsimile transmission of the SAE information is also acceptable. The fax number is +1-714-796-9504 (backup number is +1-714-246-5295).
- In rare circumstances and in the absence of facsimile equipment, notification by telephone is acceptable with a copy of the SAE form, sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE form within the designated reporting time frames.
- Contacts for SAE reporting can be found on the protocol title page.



# 10.3. Appendix 3: Abbreviations

| Abbreviation/Term | Definition |
|---|---|
| AE | adverse event |
| AESI | adverse event of special interest |
| AUC <sub>0-last,ss</sub> | area under the plasma concentration versus time curve from time 0 to the last measurable concentration, at steady state |
| bpm | beats per minute |
| C/D | cup to disc |
| CDISC | Clinical Data Interchange Standards Consortium |
| CDVA | corrected distance visual acuity |
| CFR | Code of Federal Regulations |
| $C_{min,ss}$ | minimum plasma drug concentration at steady state |
| CRF | case report form |
| DCIVA | distance-corrected intermediate visual acuity |
| DCNVA | distance-corrected near visual acuity |
| DET | dry eye test |
| eCRF | electronic case report form |
| EOS | end of the study |
| FDA | Food and Drug Administration |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| HRT | hormonal replacement therapy |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonization |
| ID | identification |
| IEC | independent ethics committee |
| IOP | intraocular pressure |
| IRB | institutional review board |
| ITT | intent-to-treat |
| IxRS | interactive electronic response system |
| LASIK | laser-assisted in situ keratomileusis |
| MMRM | mixed model repeated measure |
| NCI | National Cancer Institute |
| NEI VFQ-25 | National Eye Institute Visual Function Questionnaire 25 |
| NVPTQ | Near Vision Presbyopia Task-based Questionnaire |
| OD | right eye |
| OS | left eye |
| OSDI | Ocular Surface Disease Index |
| | L |



| Abbreviation/Term | Definition |
|-------------------|--------------------------------------------|
| PICQ | Presbyopia Impact and Coping Questionnaire |
| PK | pharmacokinetic |
| PRK | photorefractive keratectomy |
| PRO | patient reported outcomes |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SoA | schedule of activities |
| TEAE | treatment-emergent adverse event |
| VAS | visual analog scale |
| WOCBP | women of childbearing potential |



# 10.4. Appendix 4: Standard Discontinuation Criteria

| CDISC Submission Value | CDISC Definition |
|---|---|
| AE | Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. For further information, see the ICH Guideline for Clinical Safety Data Management: Definitions and Standards for Expedited Reporting (modified from ICH E2A) Synonyms: side effect, adverse experience. See also SAE, serious adverse experience. (CDISC glossary) |
| Completed | To possess every necessary or normal part or component or step; having come or been brought to a conclusion (NCI) |
| Death | The absence of life or state of being dead (NCI) |
| Lack of efficacy | The lack of expected or desired effect related to a therapy (NCI) |
| Lost to follow-up | The loss or lack of continuation of a subject to follow-up |
| Non-compliance with study drug | An indication that a subject has not agreed with or followed the instructions related to the study medication (NCI) |
| Other | Different than the one(s) previously specified or mentioned (NCI) |
| Physician decision | A position, opinion or judgment reached after consideration by a physician with reference to subject (NCI) |
| Pregnancy | Pregnancy is the state or condition of having a developing embryo or fetus in the body (uterus), after union of an ovum and spermatozoon, during the period from conception to birth. (NCI) |
| Progressive disease | A disease process that is increasing in extent or severity (NCI) |
| Protocol deviation | An event or decision that stands in contrast to the guidelines set out by the protocol (NCI) |
| Screen failure | The potential subject who does not meet one or more criteria required for participation in a trial |



| CDISC Submission Value | CDISC Definition |
|---|---|
| Site terminated by sponsor | An indication that a clinical study was stopped at a particular site by its sponsor (NCI) |
| Study terminated by sponsor | An indication that a clinical study was stopped by its sponsor (NCI) |
| Withdrawal by subject | An indication that a study participant has removed itself from the study (NCI) |



# 10.5. Appendix 5: Study Tabular Summary

| Parameter Group | Parameter | Value |
|---|---|---|
| Trial information | Trial Title | A Phase 3, Multicenter, Double-Masked,<br>Randomized, Vehicle-Controlled, Parallel-<br>Group Study Evaluating the Safety and<br>Efficacy of AGN-190584 in Participants<br>with Presbyopia |
| | Clinical Study Sponsor | Allergan, Inc. |
| | Trial Phase Classification | Phase 3 Trial |
| | Trial Indication | Presbyopia |
| | Trial Indication Type | Treatment |
| | Trial Type | Efficacy |
| | | Safety |
| | | Pharmacokinetics |
| | Trial Length | 30 days plus up to 30-day screening period |
| | Planned Country of Investigational Sites | United States |
| | Planned Number of Participants | 300 |
| | FDA-Regulated Device Study | No |
| | FDA-Regulated Drug Study | Yes |
| | Pediatric Study | No |
| Participant information | Diagnosis Group | Presbyopia |
| | Healthy Participant Indicator | No |
| | Planned Minimum Age of Participants | 40 |
| | Planned Maximum Age of Participants | 55 |
| | Sex of Participants | Male or female |
| | Stable Disease Minimum Duration | Not specified |



| Parameter Group | Parameter | Value |
|---|---|---|
| Treatments | Investigational Therapy or Treatment | AGN-190584 (Pilocarpine HCl 1.25%<br>Ophthalmic Solution) |
| | Intervention Type | Drug |
| | Pharmacological Class of Invest. Therapy | Cholinergic agonist |
| | Dose per Administration | 1 bilaterally |
| | Dose Units | Drop |
| | Dosing Frequency | Once daily |
| | Route of Administration | Topical eye drop |
| | Current Therapy or Treatment | No |
| | Added on to Existing Treatments | No |
| | Control Type | Vehicle |
| | Comparative Treatment Name | AGN-190584 Vehicle |
| Trial design | Study Type | Interventional |
| | Intervention Model | Parallel |
| | Planned Number of Arms | 2 |
| | Trial is Randomized | Yes |
| | Randomization Quotient | 1:1 |
| | Trial Blinding Schema | Double-masked |
| | Stratification Factors | Age (2 groups: ≤ 50 years and > 50 years); baseline binocular DCNVA (2 groups: 20/40 to 20/60 inclusively, and worse than 20/60); iris color (brown and non-brown), and emmetropes/non-emmetropes |
| | Adaptive Design | No |
| | Study Stop Rules | None |



# 10.6. Appendix 6: Contraceptive Guidance and Collection of Pregnancy Information

#### **Definitions:**

#### **WOCBP**

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

#### Women in the following categories are not considered WOCBP:

- 1. Premenarchal
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's: review of the participant's medical records, medical examination, or medical history interview.

#### 3. Postmenopausal female

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or HRT. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
- Females on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### **Contraception Guidance:**

#### **Female Participants**

Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception consistently and correctly as described in Table 10–1.
















































































































# 10.8. Appendix 8: Patient Reported Outcomes Questionnaires, Descriptions, and Instructions













































































#### 10.8.2. Near Vision Presbyopia Task-based Questionnaire

# **Near Vision Presbyopia Task-based Questionnaire (NVPTQ)**

**Instructions:** This questionnaire includes 12 questions on four reading tasks that you are about to complete.

You will be asked to read text from the following examples:

- Paragraph from a book
- Newspaper article
- Menu
- Nutrition label




































| $\infty$ |
|---------------|
| $\overline{}$ |
| $\circ$ |
| Ņ |
| ن |
| ĕ |
| $\Box$ |
| 5 |
| _ |
| à |
| æ |
| ~~ |
| a |
| ova |
| Ó |
| Ξ |
| ద |
| 느 |















































































#### 11. References

García-Lázaro S, Ferrer-Blasco T, Radhakrishnan H, Cervino A, Charman WN, Montes-Mico R. Visual function through 4 contact lens-based pinhole systems for presbyopia. J Cataract Refract Surg. 2012;38(5):858-865.

Holden BA, Fricke TR, Ho SM, Wong R, Schlenther G, Cronjé S, et al. Global vision impairment due to uncorrected presbyopia. Arch Ophthalmol. 2008;126:1731-1739.

Johnson L, Buckley JG, Scally AJ, Elliott DB. Multifocal spectacles increase variability in toe clearance and risk of tripping in the elderly. Invest Ophthalmol Vis Sci. 2007;48:1466-1471.

Lord SR, Dayhew J, Howland A. Multifocal glasses impair edge-contrast sensitivity and depth perception and increase the risk of falls in older people. J Am Geriatr Soc. 2002;50:1760-1766.

Moshirfar M, Desautels JD, Wallace RT, Koen N, Hoopes PC. Comparison of FDA safety and efficacy data for KAMRA and Raindrop corneal inlays. Int J Ophthalmol. 2017;10(9):1446-1451.

Pilocarpine hydrochloride ophthalmic solution 1%, 2%, and 4%. Package Insert. Fort Worth, TX: Alcon Laboratories, Inc. 2011.

Ruiz LA, Cepeda LM, Fuentes VC. Intrastromal correction of presbyopia using a femtosecond laser system. J Refract Surg. 2009;25(10):847-854.

Tomita M. Advances in Implantation Over the Years. Changes in technique have a direct correlation with decreases in a corneal inlay's removal rate. Cataract Refract Surg Today. 2015;June:67-68.

Tsai JC, Forbes M. Medical Management of Glaucoma. 3rd ed. West Islip, New York: Professional Communications, Inc.;2009.

Tucker J, Charman WN. The depth-of-focus of the human eye for Snellen letters. Am J Optom Physiol Opt. 1975;52(1):3–21.

# Approval Date: 05-Dec-2018

# **ALLERGAN**

### 1883-301-013 Protocol Amendment 1

Date (DD/MMM/YYYY)/Time (PT)

Signed by:

**Justification** 

05-Dec-2018 10:58 GMT-080

Clinical Development Approval